CLINICAL TRIAL: NCT06547476
Title: A Phase 2, Single Arm Study Investigating the Use of Chidamide and PD-1 Antibody Combination With Anlotinib in HER2-low, Unresectable and/or Metastatic Breast Cancer
Brief Title: Chidamide and PD-1 Inhibitor Plus Anlotinib for HER2-low Breast Cancer That Has Spread or Cannot be Surgically Removed
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C56
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Immune Checkpoint Inhibitors; tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat (chidamide), PD-1 inhibitor (tislelizumab), Anlotinib (Experimental)
  Interventions: Drug: Tucidinostat (chidamide), PD-1 inhibitor (tislelizumab), anlotinib

INTERVENTIONS:
Drug: Tucidinostat (chidamide), PD-1 inhibitor (tislelizumab), anlotinib — Tucidinostat (chidamide)，30mg, po., biw PD-1 inhibitor (tislelizumab), 200mg, ivgtt. d1, q3w anlotinib, 12mg, po., d1-14, q3w

SUMMARY:
This Phase II study was designed to assess the efficacy and safety of the combination of PD-1 inhibitor, Tucidinostat (chidamide), a histone deacetylase inhibitor, and anlotinib in advanced breast cancer.

Participants must have HER2-low and PD-L1 positive （CPS≥1）breast cancer that has been treated before.

Participants' cancer:

Cannot be removed by an operation Has spread to other parts of the body

ELIGIBILITY:
Inclusion Criteria:

1. Has pathologically documented breast cancer that:

   * Is unresectable or metastatic
   * Has low-HER2 expression defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested)
   * Is HR-positive
   * Has progressed on, and would no longer benefit from, endocrine therapy
   * Has been treated with 0 to 1 prior lines of chemotherapy in the recurrent or metastatic setting
   * Was never previously HER2-positive (ICH 3+ or ISH+) on prior pathology testing (per American Society of Clinical Oncology-College of American Pathologists [ASCO-CAP] guidelines)
   * PD-L1 positive （CPS≥1）
2. Has documented radiologic progression (during or after most recent treatment)
3. Has adequate archival tumor samples available or is wiling to provide fresh biopsies prior to randomization for:

   * assessment of HER2 status
   * assessment of post-treatment status
4. Has at least 1 measurable lesion per Response Evaluation Criteria In Solid Tumors 1.1
5. Has protocol-defined adequate cardiac, bone marrow, renal, hepatic and blood clotting functions
6. Male and female participants of reproductive/childbearing potential, agrees to follow instructions for method(s) of contraception and agrees to avoid preserving ova or sperm for at least 4.5 months after treatment (or longer, per locally approved labels)

Exclusion Criteria:

1. Allergies to any monoclonal antibody or tucidinostat preparation have been known, and hypersensitivity reactions of more than 3 levels have occurred
2. Previously received histone deacetylase inhibitors,or immune checkpoint inhibitor, or angiogenesis inhibitors.
3. Subjects with any active, known or suspected autoimmune disease or history of autoimmune disease.
4. Known active CNS metastases and/or carcinomatous meningitis.
5. Received a live vaccine within 4 weeks of the first dose of study medication.
6. Major surgery received or severe traumatic injury, fracture, or ulcer occurred within 4 weeks of the first dose of study medication.
7. Pregnant or lactating female.
8. Uncontrolled clinically significant systemic diseases, including active infection, unstable angina, angina occurred within 3 months,≥ NYHA II congestive heart failure, myocardial infarction occurred within 6 months, severe arrhythmia, liver, kidney, or metabolic disease.
9. Participate in other clinical trials currently or within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Time from treatment until disease progression or death

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）
Clinical Benefit Rate (CBR) | 2 years
  the total proportion of patients with Partial Response (PR), Complete Response (CR) or Stable Disease (SD) ≥6 months
Disease Control Rate （DCR） | 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and stable disease（SD）
Overall survival (OS) | 2 years
  Time from treatment until death from any cause